CLINICAL TRIAL: NCT04873479
Title: Effect of S-ketamine Anesthetic on Inflammatory Response in Septic Patients Undergoing Abdominal Surgery:a Single Center, Randomized, Controlled Trial
Brief Title: Effect of S-ketamine Anesthetic on Inflammatory Response in Septic Patients Undergoing Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of anesthesiology , Director, Chief physician, Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASLAT20210430
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Sepsis; Acute Lung Injury
Keywords: sepsis; acute lung injury; S-ketamine; Inflammation
MeSH Terms: conditions — Sepsis; Acute Lung Injury; Inflammation | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Participants in the test group received midazolam 0.05-0.1mg /kg, sufentanil 0.1-0.2ug/kg,Etomidate 0.1-0.2mg/kg, cisatracurium 0.15-0.3mg/kg, S-ketamine 0.125mg/kg (low dose) for Anesthesia induction, followed by an infusion of remifentanil 0.05-0.15ug/kg/min and S-Ketamine 0.125mg/kg/h (low dose) and continuous inhalation of sevoflurane at 2-3%.
  Interventions: Drug: S-ketamine
- control group (Other): Participants in the control group received midazolam 0.05-0.1mg /kg, sufentanil 0.2-0.3ug/kg,Etomidate 0.2-0.3mg/kg, cisatracurium 0.15-0.3mg/kg, saline 0.125ml/kg for Anesthesia induction, followed by an infusion of remifentanil 0.1-0.3ug/kg/min and saline 0.125ml/kg/h and continuous inhalation of sevoflurane at 2-3%.
  Interventions: Other: saline

INTERVENTIONS:
Drug: S-ketamine — Participants in the test group received midazolam 0.05-0.1mg /kg, sufentanil 0.1-0.2ug/kg,Etomidate 0.1-0.2mg/kg, cisatracurium 0.15-0.3mg/kg, S-ketamine 0.125mg/kg (low dose) for Anesthesia induction, followed by an infusion of remifentanil 0.05-0.15ug/kg/min and S-Ketamine 0.125mg/kg/h (low dose) and continuous inhalation of sevoflurane at 2-3%.
  Arms: test group
Other: saline — Participants in the control group received midazolam 0.05-0.1mg /kg, sufentanil 0.1-0.2ug/kg,Etomidate 0.1-0.2mg/kg, cisatracurium 0.15-0.3mg/kg, saline 0.125ml/kg for Anesthesia induction, followed by an infusion of remifentanil 0.05-0.15ug/kg/min and saline 0.125ml/kg/h and continuous inhalation of sevoflurane at 2-3%.
  Arms: control group

SUMMARY:
This study is a randomized, double-blinded, controlled design. In this study, low doses of S-ketamine were selected for surgury treatment in septic patients under general anesthesia , Meanwhile, activity of HO-1 protein , oxidative stress and inflammatory markers in serum are measured to evaluating the effects of S-ketamine Anesthetic on inflammatory response in septic patients undergoing abdominal surgury. In addition,It is very necessary to make use of the advantages of low-dose S-ketamine in anti-inflammation, and avoid the side effects of mental symptoms, so as to guide the new direction of perioperative clinical application of S-ketamine.

DETAILED DESCRIPTION:
1. Title: Effect of S-ketamine Anesthetic on Inflammatory Response in Septic Patients Undergoing Abdominal Surgery
2. Research center: Single Center
3. The Design of the study: Randomized,double-blind, Controlled Trial
4. The population of the study: The main inclusion criteria are 18 years old or above,Patients with sepsis who need surgical treatment under general anesthesia and should be transferred to ICU for further treatment after surgery
5. Sample size: Enroll 50 patients (25 patients in each group)
6. Interventions: Participants in the test group received midazolam 0.05-0.1mg /kg, sufentanil 0.1-0.2ug/kg,Etomidate 0.1-0.2mg/kg, cisatracurium 0.15-0.3mg/kg, S-ketamine 0.125mg/kg (low dose) for Anesthesia induction, followed by an infusion of remifentanil 0.05-0.15ug/kg/min and S-Ketamine 0.125mg/kg/h (low dose) and continuous inhalation of sevoflurane at 2-3%.

   while participants in the control group was the same as the test group except for received the same volume of saline instead of S-ketamine.

   Intraoperative cisatracurium and sufentanil were added according to the circumstances.Bispectral index (BIS) was used to monitor the depth of anesthesia in two groups, and the BIS value was controlled to be 40-60, and the dose was adjusted according to the depth of anesthesia.
7. The aim of the research: To investigate the effect of S-ketamine Anesthetic on Inflammatory Response in Septic Patients Undergoing Abdominal Surgery
8. Outcome# 1) Primary outcome# the incidence of postoperative pulmonary complications 2)Secondary outcome#Inflammatory indicators: leukocyte, CRP, PCT levels;Inflammatory factors: IL-6, TNF-α, CC-16,activity of HO-1;Imaging diagnosis,such as chest X-ray,ultrasound;therapies for respiratory insufficiency,such as nasal cannula,face mask,postoperative noninvasive ventilation, re-intubation with postoperative mechanical ventilation;Incidence of postoperative adverse reactions such as restlessness, delirium, salivation, nausea, vomiting, respiratory depression, dizziness, etc;Length of stay in ICU
9. The estimated duration of the study#1-2years

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis requiring surgical treatment under general anesthesia should be transferred to ICU with endotracheal intubation for further treatment after surgery
* 18≤ age ≤85, gender and nationality is not limited
* Agree to participate in this study and sign the informed consent

Exclusion Criteria:

* Declined to participate in this study
* Patients in pregnancy or with drug allergy in this study
* Patient had chronic or acute respiratory ailments
* long-term preoperative continuous ventilatory support or oxygen dependency
* Patients are now being included in another study
* In the opinion of the attending physician or researcher, there are other conditions that are not appropriate for the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative pulmonary complications | an average of 1 week
  such as pneumonia,atelectasis ,pleural effusion,respiratory insufficiency,etc

SECONDARY OUTCOMES:
Inflammatory indicators: leukocyte, CRP, PCT levels | an average of 1 day
  leukocyte, CRP, PCT levels
Inflammatory factors | an average of 1 day
  IL-6, TNF-α, CC-16,activity of HO-1
imaging diagnosis | an average of 1 week
  chest X-ray,ultrasound
therapies for respiratory insufficiency | an average of 1 week
  nasal cannula,face mask,postoperative noninvasive ventilation, re-intubation with postoperative mechanical ventilation
Incidence of postoperative adverse reactions | an average of 1 week
  such as restlessness, delirium, salivation, nausea, vomiting, respiratory depression, dizziness, etc
Length of stay in ICU | an average of 1 month
  The time from the patient's surgery to leave the ICU
Opioid consumption | an average of 1 day
  consumption of sufentanil and remifentanil

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu MD PhD, Study Chair — Tianjin Nankai Hospital
Locations (1):
- Tianjin Nankai Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trimmel H, Helbok R, Staudinger T, Jaksch W, Messerer B, Schochl H, Likar R. S(+)-ketamine : Current trends in emergency and intensive care medicine. Wien Klin Wochenschr. 2018 May;130(9-10):356-366. doi: 10.1007/s00508-017-1299-3. Epub 2018 Jan 10. PMID 29322377
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Zanos P, Moaddel R, Morris PJ, Riggs LM, Highland JN, Georgiou P, Pereira EFR, Albuquerque EX, Thomas CJ, Zarate CA Jr, Gould TD. Ketamine and Ketamine Metabolite Pharmacology: Insights into Therapeutic Mechanisms. Pharmacol Rev. 2018 Jul;70(3):621-660. doi: 10.1124/pr.117.015198. PMID 29945898
- [Background] Welters ID, Feurer MK, Preiss V, Muller M, Scholz S, Kwapisz M, Mogk M, Neuhauser C. Continuous S-(+)-ketamine administration during elective coronary artery bypass graft surgery attenuates pro-inflammatory cytokine response during and after cardiopulmonary bypass. Br J Anaesth. 2011 Feb;106(2):172-9. doi: 10.1093/bja/aeq341. Epub 2010 Dec 7. PMID 21138901